CLINICAL TRIAL: NCT00878800
Title: A Phase I/II Clinical Trial of PXD101 in Combination With Doxorubicin in Patients With Soft Tissue Sarcomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-14
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Dose Escalation: Solid Tumors; MTD: Soft Tissue Sarcomas
Keywords: Phase I/II trial; Solid tumors; Soft tissue sarcoma; PXD101; Doxorubicin
MeSH Terms: conditions — Sarcoma | interventions — belinostat; Doxorubicin

ARMS (1):
- Experimental: PXD101 and doxorubicin (BelDox) (Experimental): 5-day PXD101 IV schedule with dose escalation combined with 1 day doxorubicin dose escalation IV
  Interventions: Drug: PXD101; Drug: Doxorubicin

INTERVENTIONS:
Drug: PXD101 — Administered in combination with doxorubicin (BelDox)
  Other Names: PXD101 (Belinostat)
Drug: Doxorubicin — Administered in combination with PXD101 (BelDox)
  Other Names: Doxorubicin (Adriamycin)

SUMMARY:
Open-label, multicentre, dose-escalation Phase I/II study to evaluate safety, efficacy, pharmacodynamics, and pharmacokinetics of the combination of PXD101 with doxorubicin administered q 3 weeks in patients with advanced solid tumours. Once the Maximum Tolerable Dose has been established, up to a total of 20-40 patients with Soft Tissue Sarcoma may be enrolled at the MTD dose level to examine efficacy and safety in this specific patient population. The trial is stopped if no more than 2 responses are seen among the first 20 of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent of an IEC (Independent Ethics Committee)-approved Information consent form
2. A. For the dose escalation phase: Patients with histological or cytological confirmed solid tumours (including sarcomas), for which there is no known curative therapy B. For the MTD expansion phase: Patients with an established diagnosis of soft tissue sarcoma in need of first line chemotherapy and with measurable disease
3. Performance status (ECOG) ≤ 2
4. Life expectancy of at least 3 months
5. Age ≥ 18 years
6. Acceptable liver, renal and bone marrow function including the following:

   1. Bilirubin ≤ 1.5 times upper limit of normal (ULN)
   2. AST ([Aspartate Amino Transferase]](SGOT), ALT (SGPT) and Alkaline Phosphatase ≤ 3 times upper limit of normal (if liver metastases are present, then ≤ 5 x ULN is allowed)
   3. Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
   4. Leucocytes > 2.5 x 109/ L, neutrophils > 1.0 x 109/L, platelets > 100 x 109/L
   5. Haemoglobin > 9.0 g/dL or > 5.6 mmol/l
7. Acceptable coagulation status: PT and APTT ([activated partial thromboplastin time ]) within ≤ 1.5 times upper limit of normal or in the therapeutic range if on anticoagulation.
8. A negative pregnancy test for women of childbearing potential. For men and women of child producing potential, the use of effective contraceptive methods during the study is required
9. Serum potassium within normal range

Exclusion Criteria:

1. Treatment with investigational agents within the last 4 weeks
2. Prior anticancer therapy, within the last 3 weeks of trial dosing including chemotherapy, radiotherapy, endocrine therapy or immunotherapy
3. Co-existing active infection or any co-existing medical condition likely to interfere with trial procedures, including significant cardiovascular disease (New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable angina, congestive heart failure requiring therapy, unstable arrhythmia or a need for anti-arrhythmic therapy, or evidence of ischemia on ECG, marked baseline prolongation of QT/QTc ([corrected QT interval ]) interval, e.g., repeated demonstration of a QTc interval > 500 msec; Long QT Syndrome; the required use of concomitant medication on PXD101 infusion days that may cause Torsade de Pointes.
4. Altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
5. Concurrent second malignancy
6. History of hypersensitivity to doxorubicin
7. A. For dose escalation phase: More than two prior doses of anthracycline, more than three prior lines of chemotherapy given for metastatic disease B. For MTD expansion phase: Prior chemotherapy
8. Bowel obstruction or impending bowel obstruction
9. Known HIV positivity
10. LVEF ([left ventricular ejection fraction]) below normal range (45% by MUGA)
11. Presence of metastatic disease that, in the opinion of the investigator, would require palliative treatment within 4 weeks of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: e-mail contact via enquires@topotarget.com, Study Director — Valerio Therapeutics
Locations (3):
- Denmark (2):
  - Århus Hospital, Department of Oncology, Aarhus
  - Herlev Hospital, Department of Oncology, Herlev
- The Royal Marsden NHS Trust, Cancer Research, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: BelDox IV (600/50): PXD101 and doxorubicin: 5-day PXD101 600 mg/m² combined with doxorubicin 50 mg/m²
- Cohort 2: BelDox IV (600/75): PXD101 and doxorubicin: 5-day PXD101 600 mg/m² combined with doxorubicin 75 mg/m²
- Cohort 3: BelDox IV (800/75): PXD101 and doxorubicin: 5-day PXD101 800 mg/m² combined with doxorubicin 75 mg/m²
- Cohort 4: BelDox IV (1000/75); MTD Expansion: BelDox IV (1000/75): PXD101 and doxorubicin: 5-day PXD101 1000 mg/m² combined with doxorubicin 75 mg/m²
Period: Overall Study
Arm/Group | Cohort 1: BelDox IV (600/50) | Cohort 2: BelDox IV (600/75) | Cohort 3: BelDox IV (800/75) | Cohort 4: BelDox IV (1000/75) | MTD Expansion: BelDox IV (1000/75)
Started | 3 | 7 | 9 | 6 | 16
Completed | 0 (Mean number of cycles administered: 4.0) | 0 (Mean number of cycles administered: 4.6) | 0 (Mean number of cycles administered: 3.0) | 0 (Mean number of cycles administered: 5.3) | 0 (Mean number of cycles administered: 6.4)
Not Completed | 3 | 7 | 9 | 6 | 16
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 1
Not completed — Progressive disease | 1 | 5 | 6 | 5 | 13
Not completed — Withdrew consent | 1 | 1 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: BelDox IV (600/50): PXD101 + doxorubicin: 5-day PXD101 600 mg/m² combined with doxorubicin 50 mg/m²
- Cohort 2: BelDox IV (600/75): PXD101 + doxorubicin: 5-day PXD101 600 mg/m² combined with doxorubicin 75 mg/m²
- Cohort 3: BelDox IV (800/75): PXD101 + doxorubicin: 5-day PXD101 800 mg/m² combined with doxorubicin 75 mg/m²
- Cohort 4: BelDox IV (1000/75); MTD Expansion: BelDox IV (1000/75): PXD101 + doxorubicin: 5-day PXD101 1000 mg/m² combined with doxorubicin 75 mg/m²
- Total: Total of all reporting groups
Arm/Group | Cohort 1: BelDox IV (600/50) | Cohort 2: BelDox IV (600/75) | Cohort 3: BelDox IV (800/75) | Cohort 4: BelDox IV (1000/75) | MTD Expansion: BelDox IV (1000/75) | Total
Number analyzed (Participants) | 3 | 7 | 9 | 6 | 16 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8 | 4 | 11 | 31
  >=65 years | 0 | 2 | 1 | 2 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4 | 0 | 7 | 15
  Male | 3 | 3 | 5 | 6 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) PXD101
Description: Maximum Tolerated Dose (MTD) of PXD101treatment
Time Frame: During Cohort 1 to 4, Cycle 1 only, up to 3 weeks
Measure: Number; unit: mg/m²
Groups:
- Dose Escalation: PXD101 and doxorubicin: 5-day PXD101 600-800-1000 mg/m² combined with doxorubicin 50-75 mg/m²
Arm/Group | Dose Escalation
Number analyzed (Participants) | 25
mg/m² | 1000

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Doxorubicin
Description: Maximum Tolerated Dose (MTD) of doxorubicin
Time Frame: During Cohort 1 to 4, Cycle 1 only, up to 3 weeks
Measure: Number; unit: mg/m2
Arm/Group | Dose Escalation
Number analyzed (Participants) | 25
mg/m2 | 75

3. Secondary Outcome: Time to Response
Time Frame: Throughout study, after every 2 cycles
Population: Includes all 41 patients in the FAS population. 37 patients were censored due to no response, 23 in the Dose Escalation group and 14 in the MTD Expansion group.
Measure: Median (Full Range); unit: months
Groups:
- MTD Expansion: PXD101 and doxorubicin: 5-day PXD101 1000 mg/m² combined with doxorubicin 75 mg/m²
Arm/Group | Dose Escalation | MTD Expansion
Number analyzed (Participants) | 25 | 16
months | NA [0.3 to NA] — Median calculation not available due to only 2 responding patients | NA [1.2 to NA] — Median calculation not available due to only 2 responding patients

4. Secondary Outcome: Duration of Response
Time Frame: Throughout study, after every 2 cycles
Population: Includes only patients with response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation | MTD Expansion
Number analyzed (Participants) | 2 | 2
Months | 3.9 [3.1 to 4.8] | 7.9 [4.4 to 11.3]

5. Secondary Outcome: Time to Progression
Time Frame: Throughout study, after every 2 cycles
Population: Includes only patients with disease progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation | MTD Expansion
Number analyzed (Participants) | 18 | 15
months | 3.7 [3.0 to 5.6] | 6.0 [1.6 to 9.7]

6. Secondary Outcome: Disease Control Rate (CR or PR or SD)
Description: The disease control rate, defined as best overall response of either objective response or stable disease (CR or PR or SD) following up to 6 cycles of treatment with confirmation according to the RECIST criteria
Time Frame: Throughout study, after every 2 cycles
Population: The full-analysis set (FAS) comprises all patients enrolled in the study and receiving at least one dose of study drug, and for whom at least one tumor assessment was performed post baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation | MTD Expansion
Number analyzed (Participants) | 25 | 16
percentage of participants | 72.0 | 68.8

7. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: Dose Limiting Toxicity (DLT) of PXD101 and doxorubicin combination treatment
Time Frame: Throughout study
Measure: Number; unit: Dose limiting toxicity
Arm/Group | Dose Escalation | MTD Expansion
Number analyzed (Participants) | 25 | 16
Dose limiting toxicity | 0 | 0

8. Primary Outcome: Objective Response (CR and PR)
Description: Measured by response rate using the RECIST (Response Evaluation Criteria in Solid Tumors) response criteria (response rate: Complete Response (CR) and Partial Response (PR)) following up to 6 cycles of treatment.
Time Frame: Throughout study, after every 2 cycles
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation | MTD Expansion
Number analyzed (Participants) | 25 | 16
percentage of participants | 8 | 12.5

9. Secondary Outcome: Belinostat AUC (Time 0 to Last Measurement)
Description: Measure the AUC of belinostat alone (Day 4 values) and in the presence of doxorubicin (Day 5 values) at the Maximum Tolerated Dose level: belinostat 1000 mg/m2 and doxorubicin 75 mg/m2
Time Frame: Cycle 1, Day 4 and Day 5, pre-infusion, at end of infusion and at 5 min, 15 min, 30 min, 1 h, 2 h, 2 h and 15 min, 2 h and 30 min, 3 h, 4 h, 6 h, 8 h and 24 h post infusion
Population: The pharmacokinetic population consisted of all patients who were dosed and had evaluable pharmacokinetic data. Dose level belinostat 1000 mg/m² and belinostat 1000 mg/m² plus doxorubicin 75 mg/m² is presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Day 4 - Belinostat 1000 mg/m²: Belinostat alone
- Day 5 - Belinostat 1000 mg/m² and Doxorubicin 75 mg/m²: Belinostat combined with doxorubicin
Arm/Group | Day 4 - Belinostat 1000 mg/m² | Day 5 - Belinostat 1000 mg/m² and Doxorubicin 75 mg/m²
Number analyzed (Participants) | 21 | 19
ng*h/mL | 23100 (35.4) | 22100 (43.2)

10. Secondary Outcome: Belinostat Cmax
Description: Measure the Cmax of belinostat alone (Day 4 values) and in the presence of doxorubicin (Day 5 values) at the Maximum Tolerated Dose level: belinostat 1000 mg/m2 and doxorubicin 75 mg/m2
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Day 4 - Belinostat 1000 mg/m² | Day 5 - Belinostat 1000 mg/m² and Doxorubicin 75 mg/m²
Number analyzed (Participants) | 21 | 19
ng/mL | 41100 (35.0) | 37000 (59.1)

11. Secondary Outcome: Belinostat t½
Description: Measure the t½ of belinostat alone (Day 4 values) and in the presence of doxorubicin (Day 5 values) at the Maximum Tolerated Dose level: belinostat 1000 mg/m2 and doxorubicin 75 mg/m2
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Day 4 - Belinostat 1000 mg/m² | Day 5 - Belinostat 1000 mg/m² and Doxorubicin 75 mg/m²
Number analyzed (Participants) | 18 | 19
hours | 1.48 (71.3) | 2.13 (119.4)

ADVERSE EVENTS:
Arm/Group | Cohort 1: BelDox IV (600/50) | Cohort 2: BelDox IV (600/75) | Cohort 3: BelDox IV (800/75) | Cohort 4: BelDox IV (1000/75) | MTD Expansion: BelDox IV (1000/75)
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/7 | 5/9 | 2/6 | 10/16
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 9/9 | 6/6 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: BelDox IV (600/50) (N=3) | Cohort 2: BelDox IV (600/75) (N=7) | Cohort 3: BelDox IV (800/75) (N=9) | Cohort 4: BelDox IV (1000/75) (N=6) | MTD Expansion: BelDox IV (1000/75) (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombosis in device (General disorders) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal absecss (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bacteriaemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: BelDox IV (600/50) (N=3) | Cohort 2: BelDox IV (600/75) (N=7) | Cohort 3: BelDox IV (800/75) (N=9) | Cohort 4: BelDox IV (1000/75) (N=6) | MTD Expansion: BelDox IV (1000/75) (N=16)
Fatigue (General disorders) | 3 | 7 | 7 | 6 | 16
Mucosal inflammation (General disorders) | 0 | 3 | 2 | 3 | 12
Injection site reaction (General disorders) | 0 | 0 | 3 | 3 | 10
Pyrexia (General disorders) | 1 | 1 | 3 | 1 | 4
Pain (General disorders) | 0 | 2 | 0 | 2 | 4
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 0 | 3
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0 | 3
Chills (General disorders) | 0 | 0 | 2 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 2
Thrombosis in device (General disorders) | 1 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Catheter site swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 6 | 5 | 14
Vomiting (Gastrointestinal disorders) | 1 | 4 | 4 | 3 | 12
Constipation (Gastrointestinal disorders) | 0 | 2 | 6 | 3 | 11
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 3 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal distention (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophagal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4 | 3 | 5 | 13
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 2 | 2 | 11
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 3 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 4 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 3
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Neutrophil Count (Investigations) | 0 | 1 | 1 | 4 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 3
Blood Bilirubin (Investigations) | 0 | 0 | 1 | 0 | 1
Blood Potassium Decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood Sodium Decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Electrocardiogram Qt Prolonged (Investigations) | 0 | 2 | 0 | 0 | 0
Haemoglobin (Investigations) | 0 | 1 | 1 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Weight Decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Blood Potassium (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin (Investigations) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 3 | 2 | 10
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2 | 0
Cerebral Haematoma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Device Related Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Abdominal Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tinea Pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Soft Tissue Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 2 | 2 | 0
Flushing (Vascular disorders) | 0 | 2 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 1 | 1 | 1 | 2
Lacrimation Increased (Eye disorders) | 0 | 1 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Bladder Pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal Pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Abstains From Alcohol (Social circumstances) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less